CLINICAL TRIAL: NCT04392791
Title: Balnotherapy in SLE, the First Randomised Controlled Study
Brief Title: Does Balnotherapy Influence the Qualitiy of Life in SLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polyclinic of the Hospitaller Brothers of St. John of God, Budapest (Other)
Collaborators: University of Debrecen (Other); Szeged University (Other)
Responsible Party: Principal Investigator, Tamás Bender MD, PhD. DSC, MD, PhD. DSC Head of Phisioterapy, Polyclinic of the Hospitaller Brothers of St. John of God, Budapest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 31959-2/2017/EKU
Record Dates: First submitted 2020-05-05; First posted 2020-05-19 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: SLE
MeSH Terms: interventions — Balneology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated group (Active Comparator): The participants received thermal water therapy
  Interventions: Other: balneotherapy
- Control group (No Intervention): The participants haven't received thermal water therapy

INTERVENTIONS:
Other: balneotherapy — Balneotherapy, a medical remedy, with medically and legally recognized mineral waters for therapeutic and rehabilitation purposes
  Arms: Treated group

SUMMARY:
The aim of this study was to investigate the effects of balneotherapy on the quality of life and on work productivity of SLE patients.

DETAILED DESCRIPTION:
SLE patients in remission/low disease activity of three immunology centers were included in this randomized, controlled, follow-up study. In addition to the standard of care (SOC) sixteen out of the thirty SLE patients received balneotherapy (15 times, for 30 minutes) and fourteen patients received the SOC only. Prevalidated survey instruments including LupusQol, SF36, and WPAI questionnaires were recorded.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SLE according to SLICC/ACR, 2012 criteria;
* remission or low disease activity, evaluated with SLEDAI-2K

Exclusion Criteria:

* explorable psychiatric disease
* general contraindications to balneotherapy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Lupus Quality of Life (LupusQoL) | 10 weeks
  Considering the previous4-week period,34 items comprising eight domains, evaluates the physical health, emotional health, body image, pain, planning, fatigue, intimate relationshipsand burden to others. The scoring is made by domains, ranged from 0 (worst) to 100 (best
WPAI-Lupus is a disease specific questionnaire developed to measure work capacity and daily activity | 10 weeks
  Six questions, covering four topics records the prior 7 days impairment: absenteeism, presenteeism, overall work impairment, and activity impairment(Reilly). Evaluation is performed by domain, expressed as a percentage. A higher percentage corresponds to higher impairment, worse productivity.
The Short Form Health Survey (SF-36) | 10 weeks
  Evaluatingthe previous four weeks, it contains a total of 36 questions in 8 categories (physical activity, role limitation due to physical problems, physical pain, general health, vitality, social activity, role limitation due to emotional problems, and general mental health). Responses are rated 0-100 per topic, with 0 being the worst and 100 being the best quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Tamás Bender, MD, PhD. DSC, Principal Investigator
Locations (1):
- Polyclinic of Hospitaller Brothers of St. John of God, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No